CLINICAL TRIAL: NCT05232006
Title: Phase II Clinical Trial Aiming at Investigating the Effect of a PARP-inhibitor on Advanced Metastatic Breast Cancer in Germline PALB2 Mutations Carriers
Brief Title: PARP-inhibitor on Advanced Metastatic Breast Cancer in Germline PALB2 Mutations Carriers
Acronym: PALB2-PARPi-01
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P170929J
Record Dates: First submitted 2022-01-28; First posted 2022-02-09 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-01

CONDITIONS: Metastatic Breast Cancer in Germline-PALB2 Mutations Carriers
MeSH Terms: interventions — niraparib

STUDY DESIGN:
Intervention Model Description: Two-stage optimal Simon design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Niraparib (Experimental): PARP-inhibitor, Niraparib Dosage : starting 300 mg/day for patients with body weight ≥77kg and platelet counts ≥ 150 000/µl or 200 mg when body weight inferior to 77kg and/or platelet counts ≤ 150 000/µl and > 100 000/µl Pharmaceutical form : 100 mg capsules Posology : single dose daily Route of administration : oral Administration procedures : oral, daily single dose Duration of treatment : 12 cycles of 28 days each
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — Niraparib, once daily

SUMMARY:
The study aims at exploring the potential benefit of a PARP-inhibitor, Niraparib, in metastatic breast cancer developing in germline-PALB2 mutations carriers. This study is designed as a multicentre one-arm two-stage phase 2 clinical trial

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years
* PALB2 germline heterozygous mutation carrier, wild type BRCA1&2 (breast cancer 1&2) affected with metastatic breast cancer in first metastatic treatment line or beyond
* Histologically or cytologically confirmed breast cancer with evidence of metastatic disease.
* Triple Negative breast cancer; Patients affected with triple negative cancers should have received anthracyclines and taxanes in neo/adjuvant therapy.
* Or patients with Hormonal receptor positive (HR+)/ Human epidermal growth factor receptor 2 negative (HER2-) breast cancer, with treatment failure after a second line of therapy; Estrogen Receptor/ProgesteroneReceptor breast cancer positive patients must have received and progressed on currently recommended therapies in this indication (endocrine therapy, CDK4/6 inhibitors (adjuvant or metastatic)), or have a disease form that the treating physician believes to be inappropriate for recommended therapies in this indication.
* Prior therapy with an anthracycline and a taxane in an adjuvant setting.
* Prior platinum allowed as long as no breast cancer progression occurred on treatment or if given in adjuvant/neoadjuvant setting, at least 12 months elapsed from last dose to study entry.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Adequate bone marrow, kidney and liver function.
* Patients without visceral crisis

Exclusion Criteria:

* Patients with HER2 positive disease.
* Untreated and/or uncontrolled brain metastases.
* Patients in visceral crisis requiring chemotherapy
* Cytopenia, defined with the following thresholds: (i) Neutrophil count < 1500/mm3; Platelet count< 100 000/mm3; Hemoglobin <9g/dL
* Prior malignancy unless curatively treated and disease-free for > 5 years prior to study entry. Prior adequately treated non-melanoma skin cancer, in situ cancer of the cervix, ductal carcinoma in situ (DCIS) or stage I grade 1 endometrial cancer allowed.
* Known HIV (Human Immunodeficiency Virus) infection.
* Pregnant or breast-feeding women.
* Lack of affiliation to a social security benefit plan (as a beneficiary or assignee)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 4 months
  Complete or partial tumour response according to RECIST 1.1 criteria accounting for objective response rate in solid tumours at 4 cycles., based on the CT-Scan

SECONDARY OUTCOMES:
Progression-free survival | 12 months
  Time from inclusion to progression or death (all-cause) or last follow-up whichever occurs first
Overall survival | 12 months
  Time from inclusion to death (all-cause) or last follow-up whichever occurs first
Tumoral response | 12 months
  Partial Response or Complete Response or Stable Disease, as per to RECIST 1.1 criteria for tumoral response, based on CT-Scan
Duration of response | 12 months
  Time to treatment failure, defined as time between inclusion and treatment discontinuation (any reason: death, disease progression, toxicity) or last follow-up
Adverse event rate | 72 months
  Adverse events (clinical and biological) between inclusion and 72 months
Quality of Life variation | 12 months
  European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life C30 Questionnaire, evaluated every 3 months, from inclusion to 12 month

IPD SHARING:
Plan to Share IPD: Undecided